CLINICAL TRIAL: NCT06858553
Title: A Prospective, Multi-center Study to Characterize Intestinal Fibrosis in Patients With Crohn's Disease (CD) Using MR Enterography (MRE)-Based Artificial Intelligence
Brief Title: AI-Assisted MRE for Intestinal Fibrosis in Crohn's Disease
Status: Recruiting | Type: Observational
Sponsor: Minhu Chen (Other)
Collaborators: Sixth Affiliated Hospital, Sun Yat-sen University (Other); Sir Run Run Shaw Hospital (Other); Jinling Hospital, China (Other); MSD R&D (China) Co., Ltd. (Industry); Ruijin Hospital (Other)
Responsible Party: Sponsor-Investigator, Minhu Chen, Professor, First Affiliated Hospital, Sun Yat-Sen University
Organization: First Affiliated Hospital, Sun Yat-Sen University (Other)
Other Study IDs: No.840[2024]; MISP-102507 (Other Grant/Funding Number: MSD R&D(CHINA)CO.,LTD)
Record Dates: First submitted 2025-02-19; First posted 2025-03-05 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-08

CONDITIONS: Crohn Disease (CD)
Keywords: MRE; Artificial Intelligence; Crohn Disease; Fibrosis
MeSH Terms: conditions — Crohn Disease; Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples With DNA — Surgical bowel specimens from patients with Crohn's disease who underwent surgery due to strictures.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- training group: This group of patients is used in the training phase of the predictive model to fit an appropriate model.
- validation group: This group of patients is used to validate the trained model to determine whether the model has broad applicability.

SUMMARY:
Intestinal fibrotic strictures represent a severe complication of Crohn's disease (CD), affecting over half of the patients. Despite the continuous emergence of novel medications, effective treatment options remain scarce. Endoscopy fails to identify the full-thickness fibrosis of the bowel wall, and standardized assessment for cross-sectional imaging has yet to be established. Previous studies have demonstrated that radiomics models based on computed tomography and deep learning models exhibit commendable diagnostic capability. Thus, this project seeks to conduct a prospective multicenter study, with plans to recruit 234 CD patients requiring bowel resection from five medical centers. The aim is to develop and validate a deep learning model based on magnetic resonance enterography (MRE) to accurately characterize intestinal fibrosis.

DETAILED DESCRIPTION:
Quality Assurance Plan The registry implements a comprehensive quality assurance (QA) plan to validate data and maintain protocol adherence. This includes routine site monitoring, regular audits, and verification of data consistency. Sites participating in the registry are periodically reviewed for compliance with the established operational standards.

Data Entry and Summary Process Management will enforce access regulations to ensure only authorized personnel can enter or query data. Patient information meeting inclusion criteria will be entered into a Tencent form from the hospital's medical record system. Research assistants will supplement this form with details about intestinal surgical specimens, including condition, quantity, and storage, and summarize all specimens. Researchers will summarize the MRE imaging data for the relevant patients. No one may delete, alter, copy, print, or output confidential data without management's consent.

Verification System During patient enrollment, information collection, and specimen collection, two or more research assistants or researchers will confirm the process. Relevant information will be verified again during specimen collection, labeling, and storage. In the analysis phase, researchers will recheck the accuracy of imaging, patient information, and specimens. Management will conduct a random audit every three months to verify patient inclusion criteria and confirm specimen information accuracy.

Data Dictionary A comprehensive data dictionary is used to define each variable collected within the registry. It includes the source of the variable, coding standards and any relevant normal ranges for clinical measures. This data dictionary serves as a reference to ensure uniformity in data collection and analysis.

Standard Operating Procedures (SOPs) The registry follows established Standard Operating Procedures (SOPs) for various registry functions, including patient recruitment, data collection, management, and analysis. SOPs also cover reporting procedures for adverse events, including guidelines for data reporting and event classification. Change management processes are in place to address any amendments or updates to registry protocols.

Sample Size Assessment A statistical sample size calculation has been performed to ensure that the registry is adequately powered to detect meaningful differences or effects. This calculation takes into account the expected incidence of the event of interest, anticipated variability, and the desired statistical power. The required number of participants or participant years is specified based on the primary and secondary objectives of the study.

Plan for Missing Data The registry has a clear policy for handling missing data, including cases where data may be unavailable, uninterpretable, or missing due to inconsistencies (e.g., out-of-range results). A specific protocol is followed for imputing missing values or excluding incomplete data from analysis, ensuring the final dataset remains reliable and valid for statistical analysis.

Statistical Analysis Methods Automatic recognition and segmentation of intestinal lesions in images, based on multi-parametric MRI data and artificial intelligence models, are used to evaluate intestinal fibrosis and assist in clinical decision-making. Specifically, the process includes: performing VOI annotation to generate 3D VOI; normalizing and resampling MRE images, cropping voxel intensity and applying min-max normalization; decomposing each 3D MRE lesion image into patches, and applying 5-fold data augmentation as input to the network; developing a deep learning segmentation algorithm using the nnU-Net model for automatic recognition of intestinal lesion images, with performance evaluated using the Dice similarity coefficient; constructing a ResNet model to accurately assess different degrees of intestinal fibrosis, with output as a predicted probability between 0 and 1; collecting multi-parametric MRI data prior to model construction and extracting features not affected by intestinal inflammation; excluding relevant features during model development, retaining only those reflecting intestinal fibrosis; after model construction, grouping patients based on inflammation severity and re-evaluating the AI model's recognition capability. Through these steps and the integration of multi-omics data, molecular subtyping and related prognostic analysis of patients are achieved to assist in clinical treatment decision-making.

ELIGIBILITY:
Inclusion Criteria:

1. Patients Over 18 years old with a confirmed diagnosis of CD based on the criteria of ECCO guideline.
2. Planning to receive a bowel resection due to stricture in ileum or colon, and availability of histological specimens of resected intestinal walls matched with MRE are expected to be available.
3. Clear boundaries of the target bowel tract enable accurate semi-automatic or fully automatic intestinal segmentation

Exclusion Criteria:

1. Cannot undergo MRI examination
2. Difficult to obtain suitable tissue after surgery
3. MRE imaging is of poor quality or contains artifacts
4. The target bowel is located at the anastomosis (ie, anastomotic stricture)
5. Intestinal lesions concurrent with other diseases

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of patients from five tertiary-level IBD treatment centers located in different regions of China
Sampling Method: Non-Probability Sample
Enrollment: 234 (Estimated)
Dates: Start 2025-06-03 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
histologic inflammation score | 1 week after surgery
  Histologic evaluation of intestinal surgical specimens from enrolled patients was performed using hematoxylin and eosin (H&E) staining for the histologic inflammation score. The scoring system is graded on a 0-3 scale, with higher scores indicating a greater degree of inflammatory infiltration.
histologic fibrosis score | 1 week after surgery
  Histologic evaluation of intestinal surgical specimens from enrolled patients was performed using Masson's trichrome staining for the histologic fibrosis score. The scoring system is graded on a 0-3 scale, with higher scores indicating a greater degree of fibrosis severity.
Magnetization Transfer Ratio | 4 weeks before surgery
  All enrolled patients underwent Magnetic Resonance Enterography examinations four weeks prior to surgery. Magnetization Transfer Ratio (MTR) is calculated as MTR = [1 - (Msat / M0)] × 100, where Msat represents the signal intensity with the magnetization transfer pulse applied, and M0 represents the signal intensity without the MT pulse. To minimize individual variability, MTR is normalized using the skeletal muscle MTR, making it a reliable indicator for assessing intestinal fibrosis.
Apparent Diffusion Coefficient | 4 weeks before surgery
  All enrolled patients underwent Magnetic Resonance Enterography examinations four weeks prior to surgery. The Apparent Diffusion Coefficient (ADC) is derived from diffusion-weighted imaging (DWI) and measures the movement of water molecules in tissues, indirectly reflecting inflammation and fibrosis severity. Lower ADC values suggest restricted diffusion, which is associated with fibrosis, allowing differentiation between fibrotic and non-fibrotic bowel walls.
Percentage of Enhancement Gain | 4 weeks before surgery
  All enrolled patients underwent Magnetic Resonance Enterography examinations four weeks prior to surgery. The Percentage of Enhancement Gain is calculated using % Gain = [(WSI_7min - WSI_70s) / WSI_70s] × 100, where WSI_70s and WSI_7min are the bowel wall signal intensities at 70 seconds and 7 minutes post-contrast injection, respectively. This parameter evaluates hemodynamic changes in the bowel wall, reflecting tissue perfusion characteristics related to inflammation and fibrosis.

SECONDARY OUTCOMES:
IBD Montreal classification | 2 weeks before surgery
  The Montreal classification of Crohn's disease includes three main categories: age, disease location, and disease behavior. Age (A) is classified as ≤16 years (A1), 17-40 years (A2), and ≥40 years (A3). Disease location (L) is categorized into terminal ileum (L1), colon (L2), ileocolon (L3), and upper gastrointestinal tract (L4). Disease behavior (B) is classified as non-stricturing, non-penetrating (B1), stricturing (B2), and penetrating (B3). Additionally, perianal fistulizing disease (P) can occur in association with any of the disease behavior subtypes.
Crohn's Disease Activity Index | 2 weeks before surgery
  The Crohn's Disease Activity Index (CDAI) ranges from a minimum of 0 with no fixed maximum value. When using CDAI to assess disease status, different score thresholds are commonly applied: CDAI <150 indicates remission, while CDAI ≥150 indicates active disease. Within the active disease category, 150-220 is classified as mild activity, 221-450 as moderate activity, and >450 as severe activity.
complete blood count | 2 weeks before surgery
  Calculate the quantity and percentage of each category of serum cells.
C-reactive protein | 2 weeks before surgery
  Measure the concentration of serum C-reactive protein, expressed in mg/L.
procalcitonin | 2 weeks before surgery
  Measure the concentration of serum procalcitonin, expressed in ng/mL.
erythrocyte sedimentation rate | 2 weeks before surgery
  Measure the erythrocyte sedimentation rate of the blood，expressed in mm/h.
serum albumin | 2 weeks before surgery
  Measure the level of serum albumin, expressed in g/L.

CONTACTS AND LOCATIONS:
Overall Officials: Minhu Chen, Study Chair — First Affiliated Hospital, Sun Yat-Sen University
Locations (5):
- China (5):
  - The First Affiliated Hospital,Sun Yat-sen University, Guangzhou, Guangdong
  - Sixth Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - Jinling Hospital, Affiliated Hospital of Medical School, Nanjing University, Nanjing, Jiangsu
  - Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Huangpu, Shanghai Municipality
  - Sir Run Run Shaw Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No
In this study, we do not intend to publicly release raw patient data for the following reasons:
  1. Patient Privacy Protection: Raw data may include sensitive personal information, such as names and medical history. Public release could expose this information, violating patient privacy rights and privacy regulations.
  2. Data Security: The raw data includes medical images and clinical information, which could be misused if released. Access will be restricted to the research team to ensure data security.
  3. Ethical Considerations: Informed consent was obtained from patients with clear terms regarding data usage. They did not consent to public release of raw data, and doing so could breach the original agreement.
  4. De-identification: While de-identified data may be used, raw data that could identify patients will not be released to protect their privacy.
  5. Prevention of Data Misuse: Releasing raw data could lead to misuse by unauthorized parties.

REFERENCES:
- [Background] Li XH, Feng ST, Cao QH, Coffey JC, Baker ME, Huang L, Fang ZN, Qiu Y, Lu BL, Chen ZH, Li Y, Bettenworth D, Iacucci M, Sun CH, Ghosh S, Rieder F, Chen MH, Li ZP, Mao R. Degree of Creeping Fat Assessed by Computed Tomography Enterography is Associated with Intestinal Fibrotic Stricture in Patients with Crohn's Disease: A Potentially Novel Mesenteric Creeping Fat Index. J Crohns Colitis. 2021 Jul 5;15(7):1161-1173. doi: 10.1093/ecco-jcc/jjab005. PMID 33411893
- [Background] Li X, Zhang N, Hu C, Lin Y, Li J, Li Z, Cui E, Shi L, Zhuang X, Li J, Lu J, Wang Y, Liu R, Yuan C, Lin H, He J, Ke D, Tang S, Zou Y, He B, Sun C, Chen M, Huang B, Mao R, Feng ST. CT-based radiomics signature of visceral adipose tissue for prediction of disease progression in patients with Crohn's disease: A multicentre cohort study. EClinicalMedicine. 2022 Dec 30;56:101805. doi: 10.1016/j.eclinm.2022.101805. eCollection 2023 Feb. PMID 36618894
- [Background] Li Z, Chen Z, Zhang R, et, al. Eur J Nucl Med Mol Imaging. 2024 Feb 15.
- [Background] Du JF, Lu BL, Huang SY, Mao R, Zhang ZW, Cao QH, Chen ZH, Li SY, Qin QL, Sun CH, Feng ST, Li ZP, Huang L, Li XH. A novel identification system combining diffusion kurtosis imaging with conventional magnetic resonance imaging to assess intestinal strictures in patients with Crohn's disease. Abdom Radiol (NY). 2021 Mar;46(3):936-947. doi: 10.1007/s00261-020-02765-3. Epub 2020 Sep 22. PMID 32964274
- [Background] Zhang MC, Li XH, Huang SY, Mao R, Fang ZN, Cao QH, Zhang ZW, Yan X, Chen MH, Li ZP, Sun CH, Feng ST. IVIM with fractional perfusion as a novel biomarker for detecting and grading intestinal fibrosis in Crohn's disease. Eur Radiol. 2019 Jun;29(6):3069-3078. doi: 10.1007/s00330-018-5848-6. Epub 2018 Dec 13. PMID 30547200
- [Background] Huang SY, Li XH, Huang L, Sun CH, Fang ZN, Zhang MC, Lin JJ, Jiang MJ, Mao R, Li ZP, Zhang Z, Feng ST. T2* Mapping to characterize intestinal fibrosis in crohn's disease. J Magn Reson Imaging. 2018 Apr 17. doi: 10.1002/jmri.26022. Online ahead of print. PMID 29663577
- [Background] Li Z, Lu B, Lin J, He S, Huang L, Wang Y, Meng J, Li Z, Feng ST, Lin S, Mao R, Li XH. A Type I Collagen-Targeted MR Imaging Probe for Staging Fibrosis in Crohn's Disease. Front Mol Biosci. 2021 Nov 11;8:762355. doi: 10.3389/fmolb.2021.762355. eCollection 2021. PMID 34859052
- [Background] Li XH, Mao R, Huang SY, Fang ZN, Lu BL, Lin JJ, Xiong SS, Chen MH, Li ZP, Sun CH, Feng ST. Ability of DWI to characterize bowel fibrosis depends on the degree of bowel inflammation. Eur Radiol. 2019 May;29(5):2465-2473. doi: 10.1007/s00330-018-5860-x. Epub 2019 Jan 11. PMID 30635756
- [Background] Chen YJ, Mao R, Li XH, Cao QH, Chen ZH, Liu BX, Chen SL, Chen BL, He Y, Zeng ZR, Ben-Horin S, Rimola J, Rieder F, Xie XY, Chen MH. Real-Time Shear Wave Ultrasound Elastography Differentiates Fibrotic from Inflammatory Strictures in Patients with Crohn's Disease. Inflamm Bowel Dis. 2018 Sep 15;24(10):2183-2190. doi: 10.1093/ibd/izy115. PMID 29718309
- [Background] Li XH, Mao R, Huang SY, Sun CH, Cao QH, Fang ZN, Zhang ZW, Huang L, Lin JJ, Chen YJ, Rimola J, Rieder F, Chen MH, Feng ST, Li ZP. Characterization of Degree of Intestinal Fibrosis in Patients with Crohn Disease by Using Magnetization Transfer MR Imaging. Radiology. 2018 May;287(2):494-503. doi: 10.1148/radiol.2017171221. Epub 2018 Jan 19. PMID 29357272
- [Background] Meng J, Luo Z, Chen Z, Zhou J, Chen Z, Lu B, Zhang M, Wang Y, Yuan C, Shen X, Huang Q, Zhang Z, Ye Z, Cao Q, Zhou Z, Xu Y, Mao R, Chen M, Sun C, Li Z, Feng ST, Meng X, Huang B, Li X. Intestinal fibrosis classification in patients with Crohn's disease using CT enterography-based deep learning: comparisons with radiomics and radiologists. Eur Radiol. 2022 Dec;32(12):8692-8705. doi: 10.1007/s00330-022-08842-z. Epub 2022 May 26. PMID 35616733
- [Background] Li X, Liang D, Meng J, Zhou J, Chen Z, Huang S, Lu B, Qiu Y, Baker ME, Ye Z, Cao Q, Wang M, Yuan C, Chen Z, Feng S, Zhang Y, Iacucci M, Ghosh S, Rieder F, Sun C, Chen M, Li Z, Mao R, Huang B, Feng ST. Development and Validation of a Novel Computed-Tomography Enterography Radiomic Approach for Characterization of Intestinal Fibrosis in Crohn's Disease. Gastroenterology. 2021 Jun;160(7):2303-2316.e11. doi: 10.1053/j.gastro.2021.02.027. Epub 2021 Feb 17. PMID 33609503

DOCUMENTS (1):
  • Informed Consent Form (2024-12-17): https://cdn.clinicaltrials.gov/large-docs/53/NCT06858553/ICF_000.pdf